CLINICAL TRIAL: NCT02309957
Title: Evaluation of an Acellular Osteochondral Graft for Cartilage LEsions ("EAGLE") European Post Market Study
Brief Title: EAGLE European Post Market Study
Acronym: EAGLE
Status: Completed | Type: Observational
Sponsor: Kensey Nash Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: EAGLE EU Post Market Study
Record Dates: First submitted 2014-12-02; First posted 2014-12-05 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Acute Knee Cartilage Injury; Tear of Articular Cartilage of Knee, Current
Keywords: Knee Cartilage Repair, Osteochondral Defects, BioMatrix CRD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BioMatrix CRD: All patients will receive BioMatrix CRD to repair an articular cartilage lesion or osteochondral defect.
  Interventions: Device: BioMatrix CRD

INTERVENTIONS:
Device: BioMatrix CRD

SUMMARY:
Prospective, multi-center, non-randomized, historical controlled, post-market study of patients requiring surgical repair of a focal articular cartilage lesion or osteochondral defect in the knee.

DETAILED DESCRIPTION:
BioMatrix CRD is a CE marked device that is intended to repair focal articular cartilage lesions or osteochondral defects in the knee. BioMatrix CRD™ is a sterile, biphasic, bioresorbable scaffold designed to aid in the repair of cartilage and subchondral bone. The device serves as a scaffold for cellular and extracellular matrix ingrowth supporting the regeneration of cartilage and subchondral bone.

The purpose of this post-market study is to confirm the safety and performance of the BioMatrix CRD for its intended use. Fifty (50) patients will be enrolled at up to 10 hospitals in Europe. Patients will be followed for 2 years post-operative to examine the rate of adverse events associated with the device, track improvement in knee pain and knee function over time, and assess the quality of repair tissue.

ELIGIBILITY:
Inclusion Criteria:

* Pre-procedure KOOS Pain subscale score less than or equal to 70.
* ICRS grade 3 or 4 focal articular cartilage lesion on the medial femoral condyle, lateral femoral condyle or trochlea, which measures less than or equal to15mm in diameter.
* Cartilage lesion is amenable to treatment with a single BioMatrix CRD or an osteochondral autograft.

Exclusion Criteria:

* Previous cartilage repair procedure (i.e., microfracture, OATS, ACI) at the intended implantation site.
* Clinically significant (> 5 degrees) varus or valgus malalignment in either knee.
* Osteoarthritis in the injured knee.
* Inflammatory arthropathy
* Osteomyelitis or other active infection in either lower limb.
* Cortisone or hyaluronic acid knee injections in the past 3 months
* Body mass index greater than 35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational study of patients receiving BioMatrix CRD for surgical repair of a focal articular cartilage lesion or osteochondral defect in the knee
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Rate of Implant Failure | 24 months
  Rate of implant failure resulting in device removal and/or further surgical intervention due to a device related complication

SECONDARY OUTCOMES:
Knee Related Adverse Events | 24 months
Quality of repair tissue as assessed by magnetic resonance imaging | at 24 months
Improvement in knee pain and function as reported by patients on the Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Justus Gille, PD Dr med, Principal Investigator — University Hopsital Schleswig Holstein Campus Lübeck
Locations (6):
- Germany (3):
  - University of Schleswig-Holstein, Campus Lübeck, Lübeck
  - Technische Universität München, München
  - Klinikum der Universität Regensburg, Regensburg
- Istituto Ortopedico Rizzoli, Bologna, Italy
- Maastricht University Medical Center (MUMC+), Maastricht, Netherlands
- Robert Jones & Agnes Hunt Orthopaedic Hospital, Oswestry, United Kingdom